CLINICAL TRIAL: NCT02071615
Title: Effects of Modafinil, Caffeine and Methylphenidate on Functional Brain Activity and Cognitive Performance in Healthy Volunteers: a Randomized, Placebo-controlled, Double-blind fMRI Study
Brief Title: Effects of Modafinil, Caffeine and Methylphenidate in Healthy Volunteers
Acronym: MKM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: The Volkswagen Foundation (Other)
Responsible Party: Principal Investigator, Dimitris Repantis, Dr. med., Charite University, Berlin, Germany
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2012-003882-17; DRKS00005219 (Registry Identifier: Deutsche Register Klinischer Studien (DRKS))
Record Dates: First submitted 2014-02-15; First posted 2014-02-26 (Estimated); Last update posted 2014-04-17 (Estimated); Status verified 2014-04

CONDITIONS: Healthy
Keywords: Brain Activity
MeSH Terms: interventions — Methylphenidate; Modafinil; Caffeine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Methylphenidate and placebo (Experimental): Placebo or Methylphenidate 20 mg tablet given once by mouth
  Interventions: Drug: Methylphenidate 20 mg tablet given once by mouth; Drug: placebo
- modafinil and placebo (Experimental): placebo or modafinil 200mg tablet given once by mouth
  Interventions: Drug: modafinil 200mg tablet given once by mouth; Drug: placebo
- caffein and placebo (Experimental): placebo or caffein 200mg tablet given once by mouth
  Interventions: Drug: caffein 200mg tablet given once by mouth; Drug: placebo

INTERVENTIONS:
Drug: Methylphenidate 20 mg tablet given once by mouth — 3-arm, single-drug dosage comparison study
  Other Names: Ritalin
  Arms: Methylphenidate and placebo
Drug: modafinil 200mg tablet given once by mouth — 3-arm, single-drug dosage comparison study
  Other Names: Provigil
  Arms: modafinil and placebo
Drug: caffein 200mg tablet given once by mouth — 3-arm, single-drug dosage comparison study
  Other Names: Coffeinum
  Arms: caffein and placebo
Drug: placebo

SUMMARY:
In this study the investigators compare three stimulants to each other. The effects of these agents on cognitive performance (eg, attention and memory) and on the brain are being measured. The hypothesis is that stimulants will have a positive effect on cognitive performance.

Each study participant will receive once a placebo and once methylphenidate or modafinil or caffeine. Methylphenidate (also known as Ritalin ®) is a drug that is used in the treatment of attention deficit / hyperactivity disorder (ADHD) in children, adolescents and adults. Modafinil ( Vigil ®) is a drug used in the treatment of narcolepsy (sleeping sickness). In the study. These substances are given in the study only once and in the dosages in which is also used for the treatment of the above diseases. In the case of caffeine , the dosage corresponds to two cups of coffee.

ELIGIBILITY:
Inclusion Criteria:

* Men
* 18 - 35 years
* Written consent (according to Arzneimittelgesetz (AMG) § 40 (1) 3b)
* Good knowledge of German
* Right-handedness

Exclusion Criteria:

* Known hypersensitivity to the study medication
* All contraindications to the study medication: arrhythmia, hyperthyroidism , glaucoma , pheochromocytoma , congestive heart failure , diabetes mellitus, known liver and kidney dysfunction, vascular disease , angina, haemodynamically significant congenital heart disease , cardiomyopathy , myocardial infarction, channelopathies, arterial hypertension , cerebrovascular diseases , such as cerebral aneurysm , vascular abnormalities , including vasculitis and stroke.
* Participation in other clinical trials during or within one month prior to this clinical trial
* Medical or psychological circumstances that may endanger the proper conduct of the trial
* Existing serious somatic diseases, even if they are not covered by the contraindications according to product information
* Existing psychiatric disorders and psychiatric disorders in prehistory
* Smoker or ex-smoker for less than 5 years
* Regular caffeine consumption > 4 cups per day
* Subjects with irregular day -night rhythm (eg shift workers )
* Unwillingness to the storage and disclosure of pseudonymous data as part of the clinical trial
* Accommodation in an institution by court or administrative order (according to AMG § 40 (1) 4 )
* MRI contraindications ( eg pacemakers , metallic or electronic implants , metallic splinters , tinnitus, surgical clips )

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2013-08; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Resting state parameters of functional magnetic resonance imaging (fMRI) as a measure of brain activity | 1 hour
  The resting state parameters that will be measured are regional homogeneity (ReHo) und amplitude of low frequency fluctuation (ALFF)

SECONDARY OUTCOMES:
Performance on cognitive tests | 4 hours
  A test battery covering several cognitive domaines is being used including: digit-span-Task, dual n-back, psychomotor vigilance task, reasoning task, memory task (free recall/ recognition), mental speed task.
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Dimitris Repantis, MD, Principal Investigator — Department of Psychiatry and Psychotherapy, Charité - University
Locations (1):
- Department of Psychiatry and Psychotherapy, Charité - University, Berlin, State of Berlin, Germany